CLINICAL TRIAL: NCT03113929
Title: Quantitative MRI for Non-invasive Assessment of Severity of Alcoholic Liver Disease (ALD)
Status: Active, not recruiting | Type: Observational
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Srinivasan Dasarathy, Staff, The Cleveland Clinic
Other Study IDs: 16-1663
Record Dates: First submitted 2017-04-05; First posted 2017-04-14 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Alcoholic Liver Disease
MeSH Terms: conditions — Liver Diseases, Alcoholic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional

GROUPS / COHORTS (1):
- Alcoholic Liver Disease Patients
  Interventions: Radiation: MRI

INTERVENTIONS:
Radiation: MRI — Research MRI

SUMMARY:
The current goal in the treatment of Alcoholic Liver Disease (ALD) is to manage ALD-associated complications as there are no disease-specific therapies. Identifying disease-specific therapies to slow ALD progression is critical to improving the outcomes in these patients. Despite preclinical treatment studies in animal models that have shown promise, clinical trials in ALD patients have been limited by the absence of sensitive, quantitative methods for identifying severity and monitoring progression of liver disease. The rates of progression of liver disease in ALD are variable and difficult to predict, which makes assessments of therapies difficult. Clinical measures of hepatic or biliary disease (e.g., bilirubin, transaminases) may be normal, only mildly elevated and/or stable despite ongoing organ damage. Liver biopsies are diagnostic, but are invasive and are of limited value for longitudinal monitoring. Currently clinical imaging, including standard volumetric imaging (MRI and ultrasonography) and hepatic fibrosis assessment (e.g. Fibroscan) are also of limited utility in fully staging disease severity and monitoring progression in ALD. The absence of clinically available methods for accurately determining the severity and progression of liver disease progression in ALD has limited implementation of clinical trials using novel therapeutic agents. Development of non-invasive imaging biomarkers to assess rates of liver progression will overcome this barrier and allow for such studies to be undertaken. This study intends to perform a one-time MRI on patients with ALD to search for these biomarkers that can improve the diagnosis and treatment of ALD patients.

ELIGIBILITY:
Inclusion Criteria:

* All subjects > 18 years of age, with the clinical diagnosis of ALD and native liver will be eligible

Exclusion Criteria:

* Subjects with history of combined organ transplantation
* Presumed or biopsy-confirmed ascending cholangitis within the last 3 months
* Contraindications for MRI (e.g. pacemakers, implants/hardware that is not MRI compatible)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All subjects with a diagnosis of alcoholic liver disease that have a native liver and are at least 18 years of age are eligible to participate.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2017-07-10 (Actual); Primary Completion 2027-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
T1 relaxation time | 1 hour
  Quantification of T1 relaxation time assessed over 1 hour MRI
Hepatic fat fraction | 1 hour
  Quantification of hepatic fat fraction assessed over 1 hour MRI
ASL (Arterial spin labeling) based perfusion measurements | 1 hour
  Quantification of ASL (Arterial spin labeling) based perfusion measurement in Quantification of arterial spin labeling assessed over 1 hour MRI
Signs of portal hypertension | 1 hour
  Asses the presence or absence of splenomegaly and varices over a 1 hour MRI to help determine portal hypertension

CONTACTS AND LOCATIONS:
Locations (1):
- Cleveland Clinic Foundation, Cleveland, Ohio, United States